CLINICAL TRIAL: NCT02208479
Title: Diaphragmatic Dysfunction in Cardiac Surgery: Observational Study
Brief Title: Cardiac Surgery and Diaphragm Function
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 2014-13
Record Dates: First submitted 2014-08-01; First posted 2014-08-05 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Cardiac Surgery
Keywords: cardiac surgery; diaphragm dysfunction; mechanical ventilation weaning; respiratory paralysis; muscle weakness; cardiac bypass; valvular surgery; respiratory insufficiency
MeSH Terms: conditions — Respiratory Paralysis; Muscle Weakness; Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- cardiac surgery
  Interventions: Other: Non invasive ultrasound measurement of the diaphragm thickness during breathing

INTERVENTIONS:
Other: Non invasive ultrasound measurement of the diaphragm thickness during breathing

SUMMARY:
Diaphragm dysfunction is common after cardiac surgery and may delay weaning from mechanical ventilation and cause respiratory distress.

The investigators' main objective is to determine the incidence of diaphragm dysfunction ( using the non-invasive ultrasonic method by calculating the inspiratory diaphragmatic thickening fraction) in a selected population of cardiac surgery patients during weaning from mechanical ventilation.

The second endpoints are to determine the associated risk factors to post-operative diaphragm weakness and the consequence on the patient outcome.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old and older
* planned surgery
* ready for weaning from mechanical ventilation

Exclusion Criteria:

* protected patient
* patient refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient admitted in Intensive Care Unit (ICU) after planned cardiac surgery
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2014-06; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Diaphragm inspiratory thickening fraction | At the begining of the spontaneous breathing trial (around 4hours after surgery)

SECONDARY OUTCOMES:
Diaphragm dysfunction before surgery | the day before surgery
Severity score (Euroscore) | the day before surgery
extracorporeal circulation duration | peroperative
left ventricular ejection fraction | the day before surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Unité de Réanimation Cardio-vasculaire et Thoracique, Grenoble, France

REFERENCES:
- [Background] DiNino E, Gartman EJ, Sethi JM, McCool FD. Diaphragm ultrasound as a predictor of successful extubation from mechanical ventilation. Thorax. 2014 May;69(5):423-7. doi: 10.1136/thoraxjnl-2013-204111. Epub 2013 Dec 23. PMID 24365607
- [Background] McCool FD, Tzelepis GE. Dysfunction of the diaphragm. N Engl J Med. 2012 Mar 8;366(10):932-42. doi: 10.1056/NEJMra1007236. No abstract available. PMID 22397655
- [Background] Jaber S, Petrof BJ, Jung B, Chanques G, Berthet JP, Rabuel C, Bouyabrine H, Courouble P, Koechlin-Ramonatxo C, Sebbane M, Similowski T, Scheuermann V, Mebazaa A, Capdevila X, Mornet D, Mercier J, Lacampagne A, Philips A, Matecki S. Rapidly progressive diaphragmatic weakness and injury during mechanical ventilation in humans. Am J Respir Crit Care Med. 2011 Feb 1;183(3):364-71. doi: 10.1164/rccm.201004-0670OC. Epub 2010 Sep 2. PMID 20813887
- [Derived] Moury PH, Cuisinier A, Durand M, Bosson JL, Chavanon O, Payen JF, Jaber S, Albaladejo P. Diaphragm thickening in cardiac surgery: a perioperative prospective ultrasound study. Ann Intensive Care. 2019 Apr 24;9(1):50. doi: 10.1186/s13613-019-0521-z. PMID 31016412